CLINICAL TRIAL: NCT06989567
Title: A Phase III, Multi-Center, Double-Blind, Placebo-Controlled, Randomized Study of Intravenous L-Citrulline in Sickle Cell Disease Presenting to Emergency Departments in Acute Vaso-Occlusive Crisis in Children, Adolescents and Young Adults (6 to 21 Years)
Brief Title: A Study of Intravenous L-Citrulline in Patients Aged 6-21 Years Old With Sickle Cell Disease Presenting to Emergency Departments in Acute Vaso-Occlusive Crisis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Asklepion Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIT-SCD-003-01
Record Dates: First submitted 2025-05-08; First posted 2025-05-25 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; citrulline; Vaso-Occlusive Crisis; Pain Crisis Relief in Sickle Cell Disease; Children and Adolescents with Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The sponsor and study vendors are also blinded in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants randomized to this arm will receive a placebo intravenous (IV) treatment designed to match the appearance and administration schedule of L-citrulline. The placebo will be given as a single bolus dose followed by a continuous infusion for up to 12 hours. All participants will continue to receive standard of care pain management for sickle cell disease, consistent with the treating site's protocol and adjusted as needed based on the patient's clinical condition.
  Interventions: Other: Placebo
- L-citrulline Intravenous Treatment Arm (Experimental): Participants randomized to this arm will receive intravenous (IV) L-citrulline, a naturally occurring amino acid being investigated for its potential to treat vaso-occlusive crises (VOCs) in sickle cell disease. The study drug will be administered as a 50 mg/kg IV bolus, followed by a continuous infusion at 9 mg/kg/hour for up to 12 hours. The investigational product is provided as an isotonic solution in vials containing L-citrulline 50 mg/mL. Treatment will begin within 120 minutes of informed consent/assent and following the initial dose of opioid or ketamine, but prior to any subsequent doses. All participants will continue to receive standard-of-care (SoC) pain management per site protocol, which may be adjusted based on clinical response to study treatment.
  Interventions: Drug: L-citrulline

INTERVENTIONS:
Drug: L-citrulline — This intervention uses intravenous L-citrulline as an acute treatment for vaso-occlusive crisis (VOC) in sickle cell disease, administered as a 50 mg/kg IV bolus followed by a 9 mg/kg/hr continuous infusion. Unlike other studies that evaluate oral citrulline or chronic VOC prevention, this study focuses on real-time symptom resolution in the emergency department setting by targeting impaired nitric oxide production and vasoconstriction. The selected dosing regimen was optimized in prior studies to achieve a therapeutic plasma concentration associated with improved pain scores and reduced opioid use, distinguishing it mechanistically and clinically from other interventions.
  Arms: L-citrulline Intravenous Treatment Arm
Other: Placebo — Placebo intravenous (IV) treatment designed to match the appearance and administration schedule of L-citrulline
  Arms: Placebo

SUMMARY:
This study is being done to learn more about a possible new treatment for pain episodes (called vaso-occlusive crises or VOCs) in children, teens, and young adults with sickle cell disease (SCD). The study will include about 120 participants between the ages of 6 and 21 who come to the emergency department (ED) with a VOC.

A VOC is a painful episode that happens with no clear cause and no signs of infection or major problems with organs like the liver or kidneys.

Before joining the study, patients and their families may be asked to learn about it and give permission (called consent or assent) while at a regular clinic visit. If that hasn't happened yet, the consent/assent process will happen at the emergency department when the patient comes in for care. If the patient meets all the study requirements, they can join the treatment part of the study.

Participants will be randomly assigned (like flipping a coin) to receive either:

L-citrulline, the study drug, or A placebo, which looks the same but has no active ingredients.

Everyone has an equal chance of getting either one. The study drug is given through an IV. It starts with one larger dose, followed by a steady infusion for up to 12 hours.

All patients in the study will still receive the usual pain treatment (called standard of care), which may include opioids. However, some patients may need fewer opioids if the study treatment helps with their pain.

If any medicines are not allowed during the study, the doctor will explain this during the consent process.

Patients can go home once:

Their pain is controlled with oral (by mouth) pain medicine, They're eating and drinking well, and They've been given a personal pain management plan to use at home.

After leaving the hospital, the study team will follow up with patients by phone about 2 days later (within a 12-hour window), again around Day 7, and again around Day 30 to check how they're doing.

DETAILED DESCRIPTION:
What is Sickle Cell Disease (SCD)? Sickle cell disease is a genetic blood condition that affects red blood cells. People with SCD have a different kind of hemoglobin (called hemoglobin S) that can make red blood cells change shape. These sickle-shaped cells can block blood flow and cause painful episodes, organ damage, and other serious complications. In the U.S., about 100,000 people live with SCD, and it affects millions worldwide.

What is a VOC? A vaso-occlusive crisis (VOC) is one of the most common and painful problems in SCD. It happens when sickled red blood cells get stuck in small blood vessels, causing pain and damage. VOC is the main reason why people with SCD go to the emergency department or hospital.

Why is This Study Being Done? While there are medicines to help prevent VOCs, there are no treatments that work well to stop a VOC once it starts. That's what this study is trying to change. Researchers are testing L-citrulline, a natural substance found in the body and in some foods, to see if it can help stop a VOC in progress and reduce the need for pain medicine.

What is L-citrulline? L-citrulline is an amino acid that helps the body make nitric oxide, a substance that opens up blood vessels and improves blood flow. People with SCD often have low levels of nitric oxide, which can make VOCs worse. By giving L-citrulline through an IV, researchers hope to increase nitric oxide and relieve pain faster.

What Did Earlier Studies Show?

Earlier studies in children and teens with SCD showed that L-citrulline was:

Safe and well tolerated Most helpful at a specific dose (50 mg/kg followed by an infusion) Effective at reducing pain and lowering the need for opioid medications in some patients

The studies also showed that very high doses might not work as well. That's why the current study uses the best dose found in earlier research.

How Will This Study Work? This study will test how well L-citrulline works in the emergency room when a patient comes in with a VOC. Everyone in the study will still receive standard pain care, including opioids if needed. Some patients will also receive L-citrulline through an IV, and others will receive a placebo (a treatment that looks the same but has no active medicine). Researchers will compare how quickly the pain improves, how much medicine is needed, and how long patients stay in the hospital.

Is L-citrulline Safe? Yes, L-citrulline has been studied in many children, including those with heart conditions and SCD. It has not caused serious side effects in these studies. In fact, children with other medical problems safely take even higher doses. The most common side effect seen was temporary low blood pressure, which happened rarely and was not serious.

Why Is This Important? People with SCD deserve better options to treat pain quickly and safely. If this study shows that L-citrulline can help shorten or ease a VOC, it could lead to better care and fewer hospital stays in the future.

What is this study testing? This study is testing whether L-citrulline, given through an IV, can help treat a pain crisis (VOC) in people with sickle cell disease (SCD) more quickly and safely than standard treatment alone. The goal is to see if it reduces pain, lowers the need for pain medications like opioids, and shortens hospital stays.

Who can join?

The study includes:

Children, teens, and young adults ages 6 to 21 years Who come to the emergency department (ED) with a VOC Who do not have other causes of pain, serious infection, or organ problems

How does the study work? About 120 patients will take part in this study.

Each person will be randomly placed (like flipping a coin) into one of two groups:

One group gets L-citrulline The other group gets a placebo (a treatment that looks the same but has no active medicine) This process is double-blinded, meaning neither the patient nor the care team will know which treatment is being given.

What is the treatment? Patients receive a dose of the study drug (or placebo) within 2 hours of giving consent and before getting more IV pain medicine.

The treatment starts with a bolus dose (a quick push of medicine) followed by a continuous IV infusion for up to 12 hours.

All patients will still receive standard sickle cell pain care, but it may be adjusted depending on how well the study treatment works.

When can patients go home?

Patients may be discharged from the hospital once:

Their pain is controlled with oral pain medicine They are eating and drinking normally They have been given a personalized pain plan to manage symptoms at home

What happens after the hospital?

Patients will be followed by the study team:

At discharge About 2 days later Around Day 7 Around Day 30

Follow-up may happen by phone. The team will ask how the patient is feeling and whether they needed more care.

What will the researchers look at?

To understand how well the treatment works, the study will measure:

Pain scores How quickly the pain crisis gets better How much pain medication is used How long the hospital stay lasts How much pain interferes with daily life (using a short survey) Blood markers of inflammation and red blood cell damage

Who is watching the safety? An independent group of experts, including doctors and a statistician, will regularly review the study's progress and safety results. This group can recommend changes or even stop the study if needed to protect patients.

Why was this dose chosen?

Earlier studies in children with SCD showed that this dose of L-citrulline (50 mg/kg + 9 mg/kg/hr infusion) was:

Well tolerated (no serious side effects) Helpful in improving pain Safe, even at higher doses in other groups of children This dose was chosen based on those positive results.

When does a patient finish the study? A patient is considered to have finished the study once they complete the final visit (about 30 days after treatment).

When would the study stop early? A patient may be taken off the study if they have a serious or unexpected reaction that may be related to the treatment.

The whole study may be paused or stopped if two patients have serious reactions that the study doctor and sponsor believe may be related to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* SCD (all genotypes)
* Children, adolescents and young adults between ages 6 to 21 years
* In a steady disease state and not in the midst of any acute complication other than VOC due to SCD at study entry
* Baseline NRS score >5 or Faces Pain Scale score ≥6
* For females of childbearing potential, a negative urine pregnancy test and using an adequate method of contraception including abstinence
* Patients or parents or legal guardian of the patient who are willing and able to sign and provide consent and assent (where appropriate for the age of the child)
* Patients willing to begin study treatment within 120 minutes after providing informed consent/assent and soon after the first/initial dose, but before any subsequent doses of IV opioid or ketamine

Exclusion Criteria:

* Current pain lasting >3 days
* History of 9 hospital admissions in the prior year
* Participation in a clinical trial of a new therapy for SCD within the last 1 month
* Presence of any other complication related to SCD such as splenic sequestration, hepatic sequestration, stroke, avascular necrosis of the hip/shoulder, acute priapism, acute renal dysfunction, acute chest syndrome and other major medical conditions or organ dysfunction
* Hypotension requiring clinical intervention; hemodynamic instability; septic shock
* Severe anemia (hemoglobin <6 g/dL)
* Systemic steroid therapy within the last 24 hours
* Use of inhaled NO or medications that are known to cause hypotension (e.g., nitrates, sildenafil, tadalafil, vardenafil, osildenafil, or arginine) within the last 30 days
* Serum creatinine levels:
* Age 6-13 years: >0.9 mg/dL
* Age 14-17 years: >1.0 mg/dL
* Age ≥18 years: >1.5 mg/dL
* Report of fever (>38°C) within the last 24 hours
* Presence of acute chest syndrome, sepsis, known bacterial infection, or hemodynamic instability
* Acute mental status or neurological changes
* Acute stroke or clinical concern for stroke
* Patients with inability to have assent given (ages 6 to 17 years) or consent (ages 18 through 21 years).

Note: Parents or legal guardians can provide consent for patients who are unable to provide assent (e.g., sleepy or preoccupied by their pain).

* History of allergic reaction to L-citrulline product or dextrose
* Unreliable venous access
* The PI considers that the patient will be unable to comply with the study requirements
* Patients pre-planned for admission on arrival in ED

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Change in pain score from baseline to discharge | From enrollment to hospital discharge (typically within 12 to 72 hours), up to max of 30 day study duration
  This outcome measures the change in self-reported pain using either the Numeric Rating Scale (NRS) or the Faces Pain Scale. Participants will rate their pain at baseline (prior to study treatment) and again at the time of hospital discharge. The pain scale used depends on the participant's age and cognitive ability. A clinically meaningful improvement is defined as a reduction of ≥2 points or ≥30% from baseline.
Time to pain crisis resolution | From start of study drug infusion to discontinuation of IV opioids (within the index hospitalization), up to max of 30 day study duration
  Time (in hours) from administration of the initial bolus dose of study drug (L-citrulline or placebo) to the end of the last IV opioid dose required during the hospitalization. This endpoint reflects how quickly the participant's vaso-occlusive crisis resolves to a degree that no longer requires intravenous opioid pain medication.

SECONDARY OUTCOMES:
Duration of hospital stay | From study drug administration to hospital discharge (typically within 12 to 72 hours), up to max of 30 day study duration up to max of 30 day study duration
  Measured in hours from the time of initial bolus dose of study drug (L-citrulline or placebo) to the time the discharge order is written. This outcome assesses how long participants remain hospitalized after receiving study treatment.
Total opioid use during hospitalization | From ED registration to hospital discharge, up to max of 30 day study duration
  The total amount of opioids administered (converted to morphine-equivalent dose in mg/kg) from emergency department (ED) registration until the discharge order is written.
Proportion of patients with ≥30% reduction in opioid use | From start of study drug administration to hospital discharge, up to max of 30 day study duration
  The percentage of patients whose total opioid dose over the course of hospitalization was reduced by 30% or more compared to the dose given prior to study treatment.
Change in Patient-Reported Outcomes Measurement Information System Pain Interference Score | From baseline to Day 7 (+2) post-enrollment
  Assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form, which measures how pain affects a participant's ability to engage in daily activities on a scale from 1 to 5, with lower scores indicating lower pain interference. The change is calculated from baseline to Day 7 (+2).
Hospital admission rate | From ED presentation through hospital discharge or decision not to admit, up to max of 30 day study duration
  The percentage of participants admitted as in-patients due to sickle cell disease or complications related to vaso-occlusive crisis (VOC).

OTHER OUTCOMES:
Healthcare resource utilization | From emergency department (ED) presentation through hospital discharge, up to max of 30 day study duration
  This outcome measures differences in healthcare resource use between treatment groups, such as the number and duration of hospital admissions, procedures, and other health system interactions related to managing vaso-occlusive crisis (VOC). The analysis may include indirect estimates of healthcare savings associated with reduced admissions or shorter hospital stays.
Cost utility and cost benefit | From ED presentation through Day 30 follow-up
  This outcome evaluates the cost-effectiveness of L-citrulline versus placebo by examining costs in relation to health benefits, including quality of life. Analyses will incorporate changes in pain resolution time (pain measured using the Numeric Rating Scale (NRS) or the Faces Pain Scale) and use quality-adjusted life year (QALY) models (measured in QALY units) where applicable. Monetary valuation of hospital utilities may also be used for modeling financial impact. Composite results will be reported as a correlation between cost and effectiveness.
Change from baseline in hemoglobin concentration | From baseline to discharge and at 48 hours post-bolus dose
  This outcome assesses the change in hemoglobin concentration (g/dL) as a biomarker of hemolysis. An increase in hemoglobin levels may indicate reduced hemolysis and improved disease status.
Change from baseline in serum bilirubin concentration | From baseline to discharge and at 48 hours post-bolus dose
  This outcome evaluates the change in serum bilirubin (mg/dL), a marker of red blood cell breakdown and liver function. Decreased levels may indicate reduced hemolysis.
Change from baseline in lactate dehydrogenase (LDH) levels | From baseline to discharge and at 48 hours post-bolus dose
  This outcome evaluates the change in LDH levels (mg/dL), an indicator of cell turnover and hemolysis. A reduction in LDH may correlate with reduced disease activity.
Change from baseline in reticulocyte count | From baseline to discharge and at 48 hours post-bolus dose
  This outcome measures the change in reticulocyte count (10^9/L) to evaluate bone marrow response to hemolysis. A decrease may indicate treatment effectiveness in reducing red blood cell destruction.
Change from baseline in C-reactive protein (CRP) concentration | From baseline to discharge and at 48 hours post-bolus dose
  This outcome measures CRP levels (mg/L) as a marker of systemic inflammation. Decreased CRP may reflect reduced inflammatory activity associated with treatment.
Maximum Plasma Concentration (Cmax) of L-citrulline | From time of first dose through 6 hours post-dose, with additional samples collected at discharge or as needed, up to max of 30 day study duration
  This outcome measures the peak plasma concentration (Cmax) of L-citrulline following dosing. Cmax will be used in subsequent analyses to evaluate pharmacokinetic-pharmacodynamic relationships with clinical outcomes like symptom improvement (e.g., pain reduction or time to crisis resolution). Data will help define therapeutic exposure ranges.
Area Under the Plasma Concentration-Time Curve (AUC) for L-citrulline | From time of first dose through 6 hours post-dose, with additional samples collected at discharge or as needed, up to max of 30 day study duration
  This outcome measures AUC, a marker of overall L-citrulline exposure over time. AUC values will be evaluated in relation to clinical endpoints such as symptom improvement and time to crisis resolution. Data will help define therapeutic exposure ranges.
Steady-State Plasma Concentration (Css) of L-citrulline | From time of first dose through 6 hours post-dose, with additional samples collected at discharge or as needed, up to max of 30 day study duration
  This outcome measures steady-state plasma concentration (Css) of L-citrulline when achieved during the study. Css will define therapeutic exposure ranges.

CONTACTS AND LOCATIONS:
Overall Officials: Suvankar Majumdar, MD, Principal Investigator — Center for Cancer and Blood Disorders, Children's National Hospital
Locations (6):
- United States (6):
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of Miami, Coral Gables, Florida
  - Emory University, Atlanta, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - East Carolina (University of North Carolina), Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: No
The study protocol does not specify plans to share individual participant data outside of the sponsor and authorized research team members.

REFERENCES:
- [Background] Platt OS, Thorington BD, Brambilla DJ, Milner PF, Rosse WF, Vichinsky E, Kinney TR. Pain in sickle cell disease. Rates and risk factors. N Engl J Med. 1991 Jul 4;325(1):11-6. doi: 10.1056/NEJM199107043250103. PMID 1710777
- [Background] Davis H, Gergen PJ, Moore RM Jr. Geographic differences in mortality of young children with sickle cell disease in the United States. Public Health Rep. 1997 Jan-Feb;112(1):52-8. PMID 9018289
- [Background] Sundd P, Gladwin MT, Novelli EM. Pathophysiology of Sickle Cell Disease. Annu Rev Pathol. 2019 Jan 24;14:263-292. doi: 10.1146/annurev-pathmechdis-012418-012838. Epub 2018 Oct 17. PMID 30332562
- [Background] Niihara Y, Miller ST, Kanter J, Lanzkron S, Smith WR, Hsu LL, Gordeuk VR, Viswanathan K, Sarnaik S, Osunkwo I, Guillaume E, Sadanandan S, Sieger L, Lasky JL, Panosyan EH, Blake OA, New TN, Bellevue R, Tran LT, Razon RL, Stark CW, Neumayr LD, Vichinsky EP; Investigators of the Phase 3 Trial of l-Glutamine in Sickle Cell Disease. A Phase 3 Trial of l-Glutamine in Sickle Cell Disease. N Engl J Med. 2018 Jul 19;379(3):226-235. doi: 10.1056/NEJMoa1715971. PMID 30021096
- [Background] Barak M, Hu C, Matthews A, Fortenberry YM. Current and Future Therapeutics for Treating Patients with Sickle Cell Disease. Cells. 2024 May 16;13(10):848. doi: 10.3390/cells13100848. PMID 38786070
- [Background] Niihara Y, Zerez CR, Akiyama DS, Tanaka KR. Oral L-glutamine therapy for sickle cell anemia: I. Subjective clinical improvement and favorable change in red cell NAD redox potential. Am J Hematol. 1998 Jun;58(2):117-21. doi: 10.1002/(sici)1096-8652(199806)58:23.0.co;2-v. PMID 9625578
- [Background] Brandow AM, Panepinto JA. Hydroxyurea use in sickle cell disease: the battle with low prescription rates, poor patient compliance and fears of toxicities. Expert Rev Hematol. 2010 Jun;3(3):255-60. doi: 10.1586/ehm.10.22. No abstract available. PMID 21082977
- [Background] Lanzkron S, Carroll CP, Haywood C Jr. The burden of emergency department use for sickle-cell disease: an analysis of the national emergency department sample database. Am J Hematol. 2010 Oct;85(10):797-9. doi: 10.1002/ajh.21807. PMID 20730795
- [Background] Sickle cell disease: managing acute painful episodes in hospital: Clinical guideline. London: National Institute for Health and Care Excellence (NICE); 2012 Jun 27. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK612041/ PMID 39946515
- [Background] Hassell KL. Population estimates of sickle cell disease in the U.S. Am J Prev Med. 2010 Apr;38(4 Suppl):S512-21. doi: 10.1016/j.amepre.2009.12.022. PMID 20331952
- [Background] Ansong D, Akoto AO, Ocloo D, Ohene-Frempong K. Sickle cell disease: management options and challenges in developing countries. Mediterr J Hematol Infect Dis. 2013 Nov 4;5(1):e2013062. doi: 10.4084/MJHID.2013.062. eCollection 2013. PMID 24363877
- [Background] Powars DR, Chan LS, Hiti A, Ramicone E, Johnson C. Outcome of sickle cell anemia: a 4-decade observational study of 1056 patients. Medicine (Baltimore). 2005 Nov;84(6):363-376. doi: 10.1097/01.md.0000189089.45003.52. PMID 16267411
- [Background] Piel FB, Steinberg MH, Rees DC. Sickle Cell Disease. N Engl J Med. 2017 Apr 20;376(16):1561-1573. doi: 10.1056/NEJMra1510865. No abstract available. PMID 28423290